CLINICAL TRIAL: NCT05418114
Title: Comparison of Effect of Lignocaine Only Versus Lignocaine Plus Magnesium Sulphate as Adjuvant Perineal Pain Relief in Patients Undergoing Episiotomy.
Brief Title: Lignocaine Only Versus Lignocaine Plus Magnesium Sulphate for Pain Relief After Episiotomy.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Dr. Hamna Atta, Post Graduate Resident, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Obs/Gynae-1/HFH/RMU/16
Record Dates: First submitted 2022-02-24; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Episiotomy Wound; Pain, Procedural
MeSH Terms: conditions — Pain, Procedural | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group B (No Intervention): Patients will be given local infiltration with 9 ml (180 mg) of 2% lignocaine only.
- Group A (Active Comparator): Patients will be given local infiltration with 9 ml (180 mg) of 2% lignocaine + 1 ml (500 mg) of 50% Magnesium sulphate
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — . One group (Group A) will be given local infiltration with 9 ml (180 mg) of 2% lignocaine + 1 ml (500 mg) of 50% Magnesium sulphate. Other group (Group B) will be given local infiltration with 9 ml (180 mg) of 2% lignocaine.
  Other Names: Magnesium sulphate
  Arms: Group A

SUMMARY:
Trauma to perineal area is one of common problems faced by obstetricians affecting physical, social and mental wellbeing of patients. During labor, surgical incision to perineum (episiotomy) is done to facilitate delivery of fetus. Episiotomy is associated with complication such as hemorrhage, infection, pain and wound breakdown. Pain relief after episiotomy is primary concern of obstetrician and right of patient. Pain after delivery causes delayed mobility of patient, late initiation of breast feeding and may affect mother psychologically. Magnesium sulphate is readily available in obstetric units due to its diverse uses, wide safety margins and cost-effectiveness. Magnesium is a calcium channel blocker and noncompetitive N methyl D aspartate (NMDA) receptor antagonist with anti-nociceptive effects. Blocking of NMDA receptors inhibits central sensitization due to peripheral nociceptive stimulation. The role of magnesium has been evaluated as adjuvant for intra- and post-operative pain relief in orthopedic, gynecological, and thoracic surgeries and has established role in anesthesia and obstetrics. Lignocaine given locally does not provide adequate pain relief. There is need to find adjuvants to local anesthesia for pain relief after episiotomy. There is paucity of published data on the use of Magnesium sulphate as an adjunct to local anesthetics for episiotomy or its repair. No local study has been done in this regard.

DETAILED DESCRIPTION:
Trauma to perineal area is one of common problems faced by obstetricians affecting physical, social and mental wellbeing of patients. (Perumal D. et al. 2017) During labor, surgical incision to perineum (episiotomy) is done to facilitate delivery of fetus. (Arulkumaran S. et al 2012) Episiotomy is associated with complication such as hemorrhage, infection, pain and wound breakdown. (Sule ST et al. 2003) Pain relief after episiotomy is primary concern of obstetrician and right of patient. (Brennan F. et al. 2007) Pain after delivery causes delayed mobility of patient, late initiation of breast feeding and may affect mother psychologically.

Suturing of episiotomy is done adhering to basic surgical principles of providing good pain control. (Sultan AH et al. 2014) Traditionally local analgesia using xylocaine is being used during episiotomy and repair. Despite this patients do complain of pain in postpartum period which seems less adequate for patients. One study compared infiltration of bupivacaine and lignocaine for episiotomy and found out that patients with lignocaine had higher pain score at 2, 4, and 6 h after the repair. (Abu-Zaida A. et al. 2021) One meta-analysis also determined that pain was lower with bupivacaine compared to lignocaine after episiotomy. (Fyneface Ogan S et al. 2006) Therefore it is necessary to determine other complementary methods to provide adequate pain relief after episiotomy.

Magnesium sulphate is readily available in obstetric units due to its diverse uses, wide safety margins and cost-effectiveness. Magnesium is a calcium channel blocker and noncompetitive N methyl D aspartate (NMDA) receptor antagonist with anti-nociceptive effects. Blocking of NMDA receptors inhibits central sensitization due to peripheral nociceptive stimulation. (Akhtar MI et al. 2011) Furthermore, there are peripheral NMDA receptors in the muscles, skin, and knee joints that play a role in sensory transmission of noxious signals. The nociceptors release glutamate in response to an afferent signal that binds to NMDA receptors leading to nerve depolarization and heightened sensitivity to circulating neurotransmitters. Magnesium sulphate inhibits these receptors thus producing anti-nociceptive effect. The addition of Magnesium sulphate to local anesthetics for neuraxial anesthesia prolongs the duration of anesthesia and improves the quality of analgesia. (Abd Elsalam KA et al. 2017)

The role of magnesium has been evaluated as adjuvant for intra- and post-operative pain relief in orthopedic, gynecological, and thoracic surgeries and has established role in anesthesia and obstetrics. (Akhtar MI et al. 2011) Moreover studies have determined that subcutaneous infiltration of Magnesium sulphate with local anesthetic after caesarean section prolongs the analgesic efficacy of local anesthetic without any significant adverse effects. (Kundra S et al. 2016) One recent study comparing the effects of using local infiltration of lignocaine only and lignocaine with magnesium after episiotomy sulfate determined that patients have significant pain relief after 2 hours with combination of lignocaine and magnesium sulfate. (Garba JA et al. 2021)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant ladies undergoing vaginal birth and willing to participate in the study.

Exclusion Criteria:

* Patients not willing to participate in study.
* Patients with perineal hematoma, tear or other complications developed after episiotomy
* Patients requiring additional analgesia during treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | At episiotomy
  Numeric rating scale (NRS) for pain assessment with score of 0 as "no pain" to 10 as "worst imaginable pain" will be used to assess pain.

OTHER OUTCOMES:
Pain Assessment | 2 hours after episiotomy
  Numeric rating scale (NRS) for pain assessment with score of 0 as "no pain" to 10 as "worst imaginable pain" will be used to assess pain.
Pain Assessment | 6 hours after episiotomy
  Numeric rating scale (NRS) for pain assessment with score of 0 as "no pain" to 10 as "worst imaginable pain" will be used to assess pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hamna Atta, MBBS, Principal Investigator — Rawalpindi Medical College

IPD SHARING:
Plan to Share IPD: No